CLINICAL TRIAL: NCT00841178
Title: A Randomised Controlled Trial of the Clinical and Cost Effectiveness of Endovenous Laser Therapy in the Treatment of Varicose Veins Secondary to Isolated Sapheno-Popliteal Incompetence and Short Saphenous Reflux
Brief Title: Endovenous Laser Therapy (EVLT) for Sapheno-Popliteal Incompetence and Short Saphenous Vein (SSV) Reflux: A RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELP 2
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Venous Insufficiency; Varicose Veins
Keywords: Randomised controlled trial; Venous insufficiency; Varicose veins; Quality of Life; Clinical effectiveness; Cost effectiveness
MeSH Terms: conditions — Venous Insufficiency; Varicose Veins | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Active Comparator): Patients undergo Surgery under a general anaesthetic.
  Interventions: Procedure: Surgery
- EVLT (Experimental): Patients undergo EVLT under a local anaesthetic.
  Interventions: Procedure: EVLT

INTERVENTIONS:
Procedure: Surgery — Saphenopopliteal junction ligation, stripping of the Short Saphenous vein where possible, perforator ligation and ambulatory phlebectomy, where necessary.
  Other Names: Crossectomy
  Arms: Surgery
Procedure: EVLT — EVLT of the Short saphenous vein with perforator ligation and / or ambulatory phlebectomy as required.
  Other Names: Endovenous Laser therapy, Endovenous Laser Ablation, EVLA
  Arms: EVLT

SUMMARY:
Varicose veins are a common problem, affecting up to a third of the western adult population. Most suffer with aching, discomfort, pruritis, and muscle cramps, whilst complications include oedema, eczema, lipodermatosclerosis, ulceration, phlebitis, and bleeding. This is known to have a significant negative effect on patient's quality of life (QoL).

Surgery has been used for many years, but it is known that there is a temporary decline in QoL post-op. This was demonstrated in our pilot study. Surgery leads to painful and prolonged recovery in some patients and has the risks of infection, haematoma and nerve injury.

Recurrence rates are known to be significant. Duplex of veins post surgery has demonstrated persistent reflux in 9-29% of cases at 1 year, 13-40% at 2 years, 40% at 5 years and 60% at 34 years.

26% of NHS patients were 'very dissatisfied' with their varicose vein surgery.

Newer, less invasive treatments are being developed. It would be advantageous to find a treatment that avoided the morbidity of surgery, one that could be performed as a day-case procedure under a local anaesthetic, a treatment that could offer lower recurrence rates and allow an early return to work. These should be the aims of any new treatment for varicose veins.

Endovenous Laser Treatment (EVLT) is performed under a local anaesthetic and uses laser energy delivered into the vein to obliterate it. The vein therefore need not be tied off surgically and stripped out.

The aim of this study is to compare the clinical, cost effectiveness and safety of Surgery and EVLT.

ELIGIBILITY:
Inclusion Criteria:

* Primary, symptomatic, varicose veins
* Isolated Sapheno-popliteal (SPJ) incompetence, leading to reflux in the Short saphenous vein (SSV) on duplex ultrasound
* SSV of 4mm distally
* Ability to give informed written consent

Exclusion Criteria:

* Inability to give informed written consent
* Symptomatic or complicated varicose veins not attributable to SPJ/SSV reflux
* Evidence of deep venous reflux on duplex scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2005-10 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Generic Quality of Life - Short Form-36 | 1 Week,, 6 Weeks, 3 Months, 1 Year, 2 Years

SECONDARY OUTCOMES:
Disease Specific Quality of Life - Aberdeen Varicose Vein Questionnaire | 1 Week, 6 Weeks, 3 Months, 1 Year, 2 Years
Generic quality of life - EuroQol | 1 week, 6 weeks, 3 months, 1 year, 2 years
Venous Clinical Severity Score | 3 months, 1 year, 2 years
Visual analogue pain scores | 1 week
Return to work and normal functioning | 1 week, 6 weeks
Would undergo EVLT again if necessary | 1 week, 6 weeks, 3 months, 1 year, 2 years
Complication rates | 1 week, 6 weeks, 3 months, 1 year, 2 years
Duplex assessment | 1 week, 6 weeks, 3 months, 1 year, 2 years
Cost Effectiveness | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Chetter, MBChB, Principal Investigator — University of Hull
Locations (1):
- Hull Royal Infirmary, Hull, East Yorkshire, United Kingdom

REFERENCES:
- [Derived] Samuel N, Carradice D, Wallace T, Mekako A, Hatfield J, Chetter I. Randomized clinical trial of endovenous laser ablation versus conventional surgery for small saphenous varicose veins. Ann Surg. 2013 Mar;257(3):419-26. doi: 10.1097/SLA.0b013e318275f4e4. PMID 23160149
- [Derived] Carradice D, Mazari FA, Mekako A, Hatfield J, Allgar V, Chetter IC. Energy delivery during 810 nm endovenous laser ablation of varicose veins and post-procedural morbidity. Eur J Vasc Endovasc Surg. 2010 Sep;40(3):393-8. doi: 10.1016/j.ejvs.2010.04.010. Epub 2010 May 26. PMID 20510634
- See also: Randomized clinical trial of endovenous laser ablation versus conventional surgery for small saphenous varicose veins — https://www.ncbi.nlm.nih.gov/pubmed/23160149
- See also: A randomized clinical trial of endovenous laser ablation versus conventional surgery for small saphenous varicose veins. — https://www.ncbi.nlm.nih.gov/pubmed/25720930